CLINICAL TRIAL: NCT05560945
Title: Clinical Investigation Examining the Anticaries Efficacy of Three Dentifrices (1.5% Arginine in a Calcium Base, 8.0% Arginine in a Calcium Base, and 0.32% Sodium Fluoride in a Silica Base): a Two-year Caries Clinical Study
Brief Title: 2-year Caries Clinical Study: Arginine Fluoride-Free Toothpastes vs. NaF Toothpaste
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRO-2018-12-CAR-ARG-YPZ
Record Dates: First submitted 2022-09-27; First posted 2022-09-30 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Dental Caries
Keywords: fluoride; prevention; caries; ICDAS; DMFS; arginine
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.32% Sodium Fluoride Dentifrice Toothpaste (Active Comparator): Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Interventions: Drug: 0.32% Sodium Fluoride Dentifrice Toothpaste
- 1.5% Arginine Dentifrice Toothpaste (Experimental): Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Interventions: Drug: 1.5% Arginine Dentifrice
- 8.0% Arginine Dentifrice Toothpaste (Experimental): Whole mouth brushing with a toothpaste, 2 times/day for 2 minutes each time for the duration of the study
  Interventions: Drug: 8.0% Arginine Dentifrice

INTERVENTIONS:
Drug: 0.32% Sodium Fluoride Dentifrice Toothpaste — Toothpaste
  Arms: 0.32% Sodium Fluoride Dentifrice Toothpaste
Drug: 1.5% Arginine Dentifrice — Toothpaste
  Arms: 1.5% Arginine Dentifrice Toothpaste
Drug: 8.0% Arginine Dentifrice — Toothpaste
  Arms: 8.0% Arginine Dentifrice Toothpaste

SUMMARY:
The objective of this study is to evaluate the anticaries efficacy for three dentifrices (1.5% arginine in a calcium base, 8.0% arginine in a calcium base, and 0.32% sodium fluoride in a silica base) in a two-year caries clinical study

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form signed by parent or legal guardian to permit participation of their child in the study
* Willingness and ability to use the assigned products according to instructions, availability for all appointments and likelihood of completing the clinical trial.
* Children ages 10-14 years at baseline.
* Presence of second molars or evidence of erupting permanent molars.
* Subjects should be of good general health as evidenced by a review of the medical history.
* Presence of two or more active caries lesions (ICDAS scores of 2 or greater) and with a previous caries experience (DMFS ≥ 2). Exclusion Characteristics
* Subjects presenting with any of the criteria below will be excluded from the study:
* Presence of fixed or removable prosthetic appliance or orthodontic treatment involving more than four permanent teeth.
* Use of medication that could increase the risk of developing dental caries, i.e. medication that reduces saliva flow.
* Long-term antibiotic therapy.
* Children with cognitive and/or motor impairment.
* Severe malocclusion.
* Presence of severe caries (ICDAS 5 or 6) on five or more teeth.
* Evidence of moderate to severe periodontal disease.
* Participation in any other clinical study within the 30 days preceding the clinical study.
* History of allergies or other adverse reactions to arginine, or oral care products, or their ingredients.
* Pregnant or lactating.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6000 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the incremental subject-wise Decayed Missing Filled Surfaces score after 2 year product use. | 2 year
  the minimum score is 0, maximum score is 4/5 depending on the tooth number and a higher score represents a worse outcome
The primary efficacy endpoint will be the incremental subject-wise Decayed Missing Filled Teeth scores after two year of product use. | 2 year
  the minimum score is 0, maximum score is 4/5 depending on the tooth number and a higher score represents a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yun Po E Zhang, PhD, DDS(Hons), Study Director — Colgate Palmolive
Locations (3):
- China (3):
  - School of Stomatology, Xian Jiaotong University, Xi'an, Shaanxi
  - West China School of Stomatology, Sichuan University, Chengdu, Sichuan
  - School of Stomatology Chongqing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: No